CLINICAL TRIAL: NCT02627118
Title: Clinical Study To Elucidate The Potential Effect of Dialyzer Leaching of BPA From the Fresenius Optiflux 160NR When Compared to a Non-BPA Containing Dialyzer, the Nipro ELISIO-15H
Brief Title: Potential Effect of Dialyzer Leaching of BPA From the Fresenius Optiflux 160NR Compared to the Nipro ELISIO-15H
Acronym: bisphenol-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Nipro Medical Corporation (Industry); Dialysis Clinic, Inc. (Industry)
Responsible Party: Principal Investigator, Andre A. Kaplan, MEDICAL DIRECTOR UCONN DIALYSIS CENTER, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-156-3
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-04

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dialyzer Comparison (Experimental): 2 MONTHS OF DIALYSIS WITH THE FRESENIUS 160NR followed by 2 MONTHS OF DIALYSIS WITH THE NIPRO ELISIO-15H
  Interventions: Device: FRESENIUS 160NR; Device: NIPRO ELISIO-15H

INTERVENTIONS:
Device: FRESENIUS 160NR — 2 MONTHS OF DIALYSIS WITH THE FRESENIUS 160NR DIALYZER
Device: NIPRO ELISIO-15H — 2 MONTHS OF DIALYSIS WITH THE NIPRO ELISIO-15H DIALYZER

SUMMARY:
The aim of the study is to identify hepatic enzyme and estrogen-dependent biochemical changes that occur when dialysis patients are treated with dialyzers known to leach BPA (Bisphenol-A) into the blood, such as the commercially available Fresenius F160NR, as compared with the same chemical evaluations in patients being treated with the non BPA containing Nipro Elisio-15H dialyzer. Evaluations of patient's chemistries will be obtained prior to and after 2 months of standard dialysis treatments with each dialyzer.

DETAILED DESCRIPTION:
The investigators propose to elucidate any eventual biochemical changes, and in particular, the in vivo estrogenic activity of BPA (Bisphenol-A), when BPA is being leached into the circulation by the Fresenius 160NR dialyzer as opposed to the same biochemical changes when there is no BPA being leached, as with the non-BPA containing Nipro Elisio-15H dialyzer. The estrogen dependent biochemical end points in humans include free testosterone, sex hormone binding globulin (SHBG) and thyroid binding globulin (TBG).

ELIGIBILITY:
Inclusion Criteria:

* Male ESRD patients 18 years or older
* Stable on hemodialysis for more than 3 months
* Stable hematocrit equal to or above 29 %
* Stable vascular access
* Stable anticoagulation
* No active infection
* Able to sign informed consent and able to participate in the study
* Medically stable

Exclusion Criteria:

* Participation in another study which may interfere with the planned study
* Active infection
* Medical conditions which may interfere with the study (unstable cardiac status, chronic liver disease, active hepatitis as defined by elevated liver enzymes)
* Females (It is expected that potential changes in estrogenic activity that might be seen in patients exposed to BPA will be modest and would be masked by naturally occurring variability of estrogen activity in women at varying stages of gonadal activity (pre, post-menopausal, different points in menstrual cycle, eventual pregnancy, etc). Thus, limiting study to adult males will maximize the possibility of detecting any changes in estrogenic activity.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07-11 (Actual); Study Completion 2016-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre A Kaplan, MD, Principal Investigator — University of Connecticut

REFERENCES:
- [Background] Murakami K, Ohashi A, Hori H, Hibiya M, Shoji Y, Kunisaki M, Akita M, Yagi A, Sugiyama K, Shimozato S, Ito K, Takahashi H, Takahashi K, Yamamoto K, Kasugai M, Kawamura N, Nakai S, Hasegawa M, Tomita M, Nabeshima K, Hiki Y, Sugiyama S. Accumulation of bisphenol A in hemodialysis patients. Blood Purif. 2007;25(3):290-4. doi: 10.1159/000104869. Epub 2007 Jul 2. PMID 17622711
- [Background] Huang X, Huang J, Zhang L, Zhu Y, Li Y. A novel ERalpha-mediated reporter gene assay for screening estrogenic/antiestrogenic chemicals based on LLC-MK2 cells. Toxicol Mech Methods. 2014 Dec;24(9):627-32. doi: 10.3109/15376516.2014.945107. Epub 2014 Sep 26. PMID 25045971
- [Background] Welshons WV, Nagel SC, vom Saal FS. Large effects from small exposures. III. Endocrine mechanisms mediating effects of bisphenol A at levels of human exposure. Endocrinology. 2006 Jun;147(6 Suppl):S56-69. doi: 10.1210/en.2005-1159. Epub 2006 May 11. PMID 16690810
- [Background] Lang IA, Galloway TS, Scarlett A, Henley WE, Depledge M, Wallace RB, Melzer D. Association of urinary bisphenol A concentration with medical disorders and laboratory abnormalities in adults. JAMA. 2008 Sep 17;300(11):1303-10. doi: 10.1001/jama.300.11.1303. Epub 2008 Sep 16. PMID 18799442
- [Background] Trasande L, Attina TM, Trachtman H. Bisphenol A exposure is associated with low-grade urinary albumin excretion in children of the United States. Kidney Int. 2013 Apr;83(4):741-8. doi: 10.1038/ki.2012.422. Epub 2013 Jan 9. PMID 23302717

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dialyzer Comparison
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dialyzer Comparison
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic/Latino | 3
  Hispanic | 5
  African American | 1
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: BPA Level Following 2 Months of Dialysis
Description: blood sampling of BPA (Bisphenol-A) in ng/mL following 2 months of dialysis with the Fresenius 160NR or the Nipro Elisio 15-H
Time Frame: 2 MONTHS OF TREATMENT
Population: When data was collected, BPA level was not measureable in one patient (lab reported the presence of unidentified "interfering substance") and that patient's data was removed from final analysis.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Dialyzer Comparison
Number analyzed (Participants) | 9
ng/mL
  following Fresenius 160NR dialyzer | 9.76 (14.65)
  following 2 months of Nipro Elisio 15-H dialyzer | 1.55 (1.90)
Statistical Analysis 1: Comparison: Dialyzer Comparison; Test type: Other; p = 0.05, t-test, 1 sided

ADVERSE EVENTS:
Groups:
- FRESENIUS OPTIFLUX 160NR: 2 MONTHS OF DIALYSIS WITH THE FRESENIUS OPTIFLUX 160NR
- NIPRO ELISIO-15H: 2 MONTHS OF DIALYSIS WITH THE NIPRO ELISIO-15H
Arm/Group | FRESENIUS OPTIFLUX 160NR | NIPRO ELISIO-15H
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No